CLINICAL TRIAL: NCT00010075
Title: Study Of The Survival Without Degradation To The Quality Of Life During Chemotherapy For Metastatic Breast Cancer In Women
Brief Title: Combination Chemotherapy in Treating Older Women With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068439; FRE-GERCOR-SAM-S99-1; EU-20028
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2003-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Leucovorin; Mitoxantrone

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating older women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the survival without degradation of quality of life in elderly women with metastatic breast cancer treated with leucovorin calcium, fluorouracil, and mitoxantrone.
* Determine the efficacy of this regimen, in terms of response and survival without progression, in these patients.
* Determine the tolerance of these patients to this regimen.

OUTLINE: This is a multicenter study.

Patients receive mitoxantrone IV and leucovorin calcium IV over 2 hours on day 1. Patients then receive fluorouracil IV over 46 hours on days 1-2. Treatment repeats every 21 days for a maximum of 8 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, after 3 courses, and at treatment completion.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 39 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic adenocarcinoma of the breast
* Bidimensionally measurable or evaluable disease

  * At least one non-irradiated lesion that is at least 2 cm in the greater diameter OR
  * Serous drainage, cutaneous metastasis, osseous metastasis, etc.
* No symptomatic cerebral metastasis
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 75 to 90

Sex:

* Female

Menopausal status:

* Postmenopausal

Performance status:

* WHO 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Platelet count at least 100,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3

Hepatic:

* Alkaline phosphatase less than 3 times normal
* Bilirubin less than 1.5 times normal
* Transaminases less than 3 times normal
* Total protein greater than 60%
* Albumin greater than 30 g/L

Renal:

* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* LVEF greater than 50% by echocardiogram or scintigraph
* ECG normal
* No uncontrolled angina
* No myocardial infarction within past 6 months

Other:

* No other medical illness or condition that would preclude study
* No other prior malignancy except basal cell skin cancer or curatively treated carcinoma in situ of the cervix
* No psychological, social, familial, or geographical reasons that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior adjuvant chemotherapy allowed
* No prior adjuvant anthracyclines
* No prior chemotherapy for metastatic disease

Endocrine therapy:

* One or two prior regimens of hormonal therapy allowed for metastatic disease

Radiotherapy:

* No prior radiotherapy for metastatic disease

Surgery:

* Not specified

Other:

* No concurrent participation in another study

Ages: 75 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Carola, MD, Study Chair — C.H. Senlis
Locations (6):
- France (6):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Polyclinique De Courlancy, Metz
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - C.H. Senlis, Senlis
  - Centre Medico-Chirurgical Foch, Suresnes